CLINICAL TRIAL: NCT00448864
Title: KALAHARI-1: Kallikrein Antagonist (DX-88 [Ecallantide]) Effect on Blood Loss Associated With Heart Surgery Requiring Institution of Bypass
Brief Title: Efficacy Study of Recombinant Protein (Ecallantide) to Reduce Blood Loss During Primary Coronary Bypass Grafting or Valve Repair/Replacement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Experience gained from this study is sufficient to design and facilitate the follow-on study.
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1501-001; DX-88/16 (Other: Cubist Study Number)
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — ecallantide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ecallantide - Low Dose Regimen (Experimental): Participants received a maximum of 15 milligrams (mg) ecallantide in stages. Intravenous (IV) infusion of 0.6 milligrams per milliliter (mg/mL) ecallantide was administered at 2.92 milliliters per minute (mL/min) for 20 minutes. The infusion rate was then reduced to 0.583 mL/min for 160 minutes, or until the end of cardiopulmonary bypass (CPB), whichever came first. At the termination of the initial infusion, a second infusion of 0.4 mg/mL ecallantide was started at 38 milliliters per hour (mL/hr) for 4 hours.
  Interventions: Drug: Ecallantide
- Ecallantide - High Dose Regimen (Experimental): Participants received a maximum of 91 mg ecallantide in stages. IV infusion of 0.6 mg/mL ecallantide was administered at 2.92 mL/min for 20 minutes. The infusion rate was then reduced to 0.583 mL/min for 160 minutes, or until the end of CPB, whichever came first. At the termination of the initial infusion, an infusion of normal saline was started at 38 milliliters per hour (mL/hr) for 4 hours.
  Interventions: Drug: Ecallantide
- Placebo (Placebo Comparator): Participants received placebo in stages. IV infusion placebo was administered at 2.92 mL/min for 20 minutes. The infusion rate was then reduced to 0.583 mL/min for 160 minutes, or until the end of CPB, whichever came first. At the termination of the initial infusion, a second infusion of placebo was started at 38 mL/hr for 4 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ecallantide
  Other Names: DX-88
  Arms: Ecallantide - High Dose Regimen; Ecallantide - Low Dose Regimen
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study was to assess the efficacy and safety of 2 dose levels of ecallantide versus placebo in reducing blood loss following cardiopulmonary bypass (CPB), as measured by chest tube drainage during the first 12 hours postoperatively or until the chest tube was removed, whichever came first, in patients undergoing primary coronary artery bypass grafting (CABG), single valve repair, or single valve replacement.

The secondary objective was to compare the efficacy of all ecallantide-treated participants (pooled high and low-doses) to placebo and to compare the high-dose to the low-dose ecallantide group. Other secondary objectives were to evaluate pharmacokinetics and antibody formation.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, double-blind, placebo-controlled, multi-center study designed to assess the efficacy and safety of 2 dose levels of ecallantide compared to placebo in reducing chest tube drainage in participants requiring CPB for primary CABG, single valve repair, or single valve replacement. Participants were randomized in a 3:3:2 ratio to ecallantide high-dose regimen (maximum 91 mg), ecallantide low-dose regimen (maximum 15 mg), or placebo. Randomization was stratified by surgical procedure so that participants undergoing valve replacement would be evenly distributed across treatment arms. Each participant received active drug or placebo administered in stages on the day of the surgical procedure after induction of anesthesia (Day 1).

Participants were screened up to 14 days prior to surgery. Additional study procedures were conducted on Day -1 or 1, peri-operatively, during the immediate postoperative period, and on Days 2, 4, and 7 (or at the time of discharge from the hospital), and between Days 28 and 43 (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 to ≤85 years of age
* Elective primary coronary artery bypass grafting (CABG), single valve repair, or single valve replacement requiring CPB and full sternotomy
* No plan to use desmopressin acetate (DDAVP), atrial natriuretic hormone, E-aminocaproic acid (EACA), tranexamic acid, or aprotinin during or postoperatively
* Female participants must be non-lactating and not pregnant
* If of childbearing potential, female participants must agree to use adequate contraception for 1 month after receiving study drug

Exclusion Criteria:

* Concomitant surgery including but not limited to atrial septal defect repair, multiple valve replacement, carotid endarterectomy, and combined CABG and valve procedure
* Planned hypothermic CPB using temperatures less than 28 degrees Celsius
* Weight <55 kilograms (kg)
* Major end organ dysfunction, defined as:

  * Cardiac:

    * Left ventricular ejection fraction (LVEF) < 30% by left ventriculography, echocardiogram, or catheterization (within 90 days prior to screening)
    * Use of positive IV inotropic agents within 12 hours prior to surgery
    * Preoperative use of intra-aortic balloon pump (IABP), left ventricular assist device (LVAD), or extracorporeal membrane oxygenation (ECMO)
  * Renal: Serum creatinine > 1.5 milligrams per deciliter (mg/dL)
  * Hepatic: Aspartate aminotransferase (AST) or alanine transferase (ALT) > 2.5 x upper limit normal
  * Hematologic:

    * Preoperative hematocrit (Hct) < 30%
    * Platelet count < 100,000/mm^3
    * Planned transfusion during surgical procedure
    * History or family history of bleeding or clotting disorder (for example, von Willebrand's Disease, idiopathic thrombocytopenia purpura (ITP), thrombotic thrombocytopenia purpura (TTP), hematologic malignancy)
    * Prothrombin time (PT) or activated partial thromboplastin time
    * (aPTT) > 1.5 x normal range; if receiving unfractionated heparin preoperatively, then abnormal preoperative PT/aPTT permitted
* Serious intercurrent illness or active infection
* Previous exposure to ecallantide
* Known allergy to ecallantide or any of its components, fentanyl, midazolam, isoflurane, propofol, morphine, heparin, or protamine
* Autologous blood donation ≤ 30 days month prior to surgery
* Known substance abuse within 6 months prior to surgery
* Receipt of an investigational drug or device within 30 days prior to participation in the current study
* Administration of:

  * Eptifibatide < 12 hours prior to surgery
  * Tirofiban hydrochloride (HCl) < 12 hours prior to surgery
  * Enoxaparin sodium or other low- molecular-weight heparin < 24 hours prior to surgery
  * Clopidogrel <5 days prior to surgery
  * Warfarin <5 days prior to surgery (Warfarin must be discontinued 5 days prior to surgery and PT must be < 18 seconds)
  * Ticlopidine <7 days prior to surgery
  * Abciximab <24 hours prior to surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2008-07-01 (Actual); Study Completion 2008-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Sternlicht, MD, Study Director — Dyax Corp.
Locations (15):
- United States (15):
  - St. Vincent's Hospital, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Texas Heart Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Ecallantide - High Dose Regimen: Participants received a maximum of 91 mg ecallantide in stages. IV infusion of 0.6 mg/mL ecallantide was administered at 2.92 mL/min for 20 minutes. The infusion rate was then reduced to 0.583 mL/min for 160 minutes, or until the end of CPB, whichever came first. At the termination of the initial infusion, an infusion of normal saline was started at 38 mL/hr for 4 hours.
Period: Overall Study
Arm/Group | Ecallantide - Low Dose Regimen | Ecallantide - High Dose Regimen | Placebo
Started | 27 | 29 | 19
Received at Least 1 Dose of Study Drug | 26 | 25 | 18
Started Post-operative Period | 26 | 25 | 18
Completed Post-operative Period | 26 | 25 | 18
Completed | 22 | 24 | 18
Not Completed | 5 | 5 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug.
Groups:
- Ecallantide - Low Dose Regimen: Participants received a maximum of 15 mg ecallantide in stages. IV infusion of 0.6 mg/mL ecallantide was administered at 2.92 mL/min for 20 minutes. The infusion rate was then reduced to 0.583 mL/min for 160 minutes, or until the end of CPB, whichever came first. At the termination of the initial infusion, a second infusion of 0.4 mg/mL ecallantide was started at 38 mL/hr for 4 hours.
- Total: Total of all reporting groups
Arm/Group | Ecallantide - Low Dose Regimen | Ecallantide - High Dose Regimen | Placebo | Total
Number analyzed (Participants) | 26 | 25 | 18 | 69
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 0 | 0 | 0
  BTWN | 17 | 16 | 11 | 44
  GTE65 | 9 | 9 | 7 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 3 | 14
  Male | 22 | 18 | 15 | 55

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Chest Tube Drainage During the First 12 Hours Postoperatively
Description: Mean volume of chest tube drainage during the first 12 hours postoperatively or until chest tube removal, whichever occurred first, is presented for each treatment group.
Time Frame: Up to 12 hours post admission to intensive care unit (ICU)
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Milliliters
Groups:
- Ecallantide - Low Dose Regimen: Participants received a maximum of 15 mg ecallantide in stages. Intravenous (IV) infusion of 0.6 mg/mL ecallantide was administered at 2.92 mL/min for 20 minutes. The infusion rate was then reduced to 0.583 mL/min for 160 minutes, or until the end of CPB, whichever came first. At the termination of the initial infusion, a second infusion of 0.4 mg/mL ecallantide was started at 38 mL/hr for 4 hours.
Arm/Group | Ecallantide - Low Dose Regimen | Ecallantide - High Dose Regimen | Placebo
Number analyzed (Participants) | 26 | 25 | 18
Milliliters | 729.9 (432.03) | 935.8 (510.18) | 1400.7 (1371.65)

2. Secondary Outcome: Cumulative Chest Tube Drainage at 24 Hours Postoperatively
Description: Mean volume of chest tube drainage during the first 24 hours postoperatively or until chest tube removal, whichever occurred first, is presented for each treatment group.
Time Frame: Up to 24 hours post admission to ICU
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Ecallantide - Low Dose Regimen | Ecallantide - High Dose Regimen | Placebo
Number analyzed (Participants) | 26 | 25 | 18
Milliliters | 82.9 (74.99) | 149.8 (132.27) | 225.3 (453.60)

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: up to 28 days post admission to ICU
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ecallantide - Low Dose Regimen | Ecallantide - High Dose Regimen | Placebo
Number analyzed (Participants) | 26 | 25 | 18
participants | 25 | 23 | 18

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve
Description: Results are reported in terms of the Area Under Plasma Concentration Time Curve (AUC), measured as milligram hour per liter (mg*h/L)
Time Frame: 1, 2, 4, and 8 hours after end of study drug infusion
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg*h/L
Groups:
- Ecallantide - Low Dose Regimen: Participants received a maximum of 15 milligrams (mg) ecallantide in stages. Intravenous (IV) infusion of 0.6 milligrams per milliliter (mg/mL) ecallantide was administered at 2.92 milliliters per minute (mL/min) for 20 minutes. The infusion rate was then reduced to 0.583 mL/min for 160 minutes, or until the end of cardiopulmonary bypass (CPB), whichever came first. At the termination of the initial infusion, a second infusion of 0.4 mg/mL ecallantide was started at 38 mL/hr for 4 hours.
Arm/Group | Ecallantide - Low Dose Regimen | Ecallantide - High Dose Regimen
Number analyzed (Participants) | 26 | 25
mg*h/L | 1.39 (0.589) | 13.6 (3.58)

ADVERSE EVENTS:
Arm/Group | Ecallantide - Low Dose Regimen | Ecallantide - High Dose Regimen | Placebo
Serious Adverse Events (participants affected / at risk) | 9/26 | 4/25 | 7/18
Other Adverse Events (participants affected / at risk) | 25/26 | 23/25 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecallantide - Low Dose Regimen (N=26) | Ecallantide - High Dose Regimen (N=25) | Placebo (N=18)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) — Resulted in one death
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecallantide - Low Dose Regimen (N=26) | Ecallantide - High Dose Regimen (N=25) | Placebo (N=18)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 6 (6) | 6 (6)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 5 (6) | 7 (10)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Bundle branch block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 5 (5) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal vascular thrombosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (6) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Crepitations (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Infusion site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 2 (2) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 3 (3)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 3 (3)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 9 (9) | 5 (5)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood chloride increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 3 (3) | 1 (3) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac enzymes increased (Investigations) | 3 (3) | 1 (1) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram (Investigations) | 1 (2) | 0 (0) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Mean arterial pressure decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Oxygen saturation normal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Thoracic cavity drainage test abnormal (Investigations) | 3 (3) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 3 (3)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrolyte depletion (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Staring (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 6 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Oxygen supplementation (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 7 (8) | 7 (9) | 5 (6)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other